CLINICAL TRIAL: NCT05190705
Title: A Phase II Study Evaluating Loncastuximab Tesirine in Patients With Previously Treated Waldenström Macroglobulinemia
Brief Title: Loncastuximab Tesirine in WM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shayna Sarosiek, MD (Other)
Collaborators: ADC Therapeutics S.A. (Industry)
Responsible Party: Sponsor-Investigator, Shayna Sarosiek, MD, Principal Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-622
Record Dates: First submitted 2021-12-29; First posted 2022-01-13 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Waldenstrom Macroglobulinemia
Keywords: Waldenstrom Macroglobulinemia
MeSH Terms: conditions — Waldenstrom Macroglobulinemia | interventions — loncastuximab tesirine; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Loncastuximab Tesirine + Dexamethasone (Experimental): Participants will be given
  * Loncastuximab Tesirine on Day 1 of every 28 day study cycle and continue for up to 6 cycles.
  Participants will also receive pre-medications to reduce the chance of having a sensitivity reaction to the study treatment. Participants who tolerate the study treatment without a reaction may have pre-medications changed per determination of their doctor.
  * Dexamethasone will be given prior to study treatment on Day -1 or up to 2 hours prior to loncastuximab tesirine and the day after treatment
  Interventions: Drug: Loncastuximab Tesirine; Drug: Dexamethasone

INTERVENTIONS:
Drug: Loncastuximab Tesirine — Administered by intravenous infusion
  Other Names: Zynlonta
Drug: Dexamethasone — Taken orally or administered by intravenous infusion
  Other Names: Decadron; Dexamethasone Intensol; Dexpak; Taperpak

SUMMARY:
This study is being done to examine the safety and effectiveness of loncastuximab tesirine as a possible treatment for participants with Waldenström Macroglobulinemia (WM).

The name of the study drug involved in this study is:

* Loncastuximab tesirine

DETAILED DESCRIPTION:
This is a single-arm, open-label, phase II study to evaluate the safety and efficacy of loncastuximab tesirine in patients with Waldenström Macroglobulinemia (WM) who have received at least 2 prior treatments, including an anti-CD20 antibody such as rituximab and a BTK inhibitor such as ibrutinib.

The U.S. Food and Drug Administration (FDA) has not approved loncastuximab tesirine for Macroglobulinemia (WM) but it has been approved for other uses. Loncastuximab tesirine is a type of therapy called an antibody drug conjugate. This type of treatment is an antibody to CD19, a protein that is typically found on B-cells and plasma cells in patients with Macroglobulinemia (WM). This is a targeted therapy that uses an antibody (immunoglobulin) to deliver a toxin directly to the cancer.

The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits.

It is expected that about 36 people will take part in this research study.

ADC Therapeutics is supporting this research study by providing funding and the study drug.

ELIGIBILITY:
Inclusion Criteria:

* Clinicopathological diagnosis of Waldenström Macroglobulinemia
* Symptomatic disease meeting criteria for treatment using consensus panel criteria from the Second International Workshop on Waldenström macroglobulinemia.
* At least 2 prior lines of treatment, including an anti-CD20 monoclonal antibody-containing regimen and a BTK inhibitor.
* Age 18 years or older
* Measurable disease, defined as presence of immunoglobulin M (IgM) paraprotein with a minimum serum IgM level of > 2 times the upper limit normal.
* ECOG performance status ≤2 (Karnofsky ≥60%, see Appendix A)
* Women of childbearing potential: Females of childbearing potential (FCBP) must agree to use two reliable forms of contraception simultaneously or have or will have complete abstinence from heterosexual intercourse during the following time periods related to this study: 1) while participating in the study; and 2) for at least 9 months after discontinuation from the study. FCBP must be referred to a qualified provider of contraceptive methods if needed.
* Men must agree to use a latex condom during sexual contact with a female of childbearing potential (FCBP) even if they have had a successful vasectomy 1) while participating in the study; and 2) for at least 6 months after discontinuation from the study.
* Participants must have normal organ and marrow function as defined below:

  * Absolute neutrophil count ≥1000/ uL. Growth factors are not permitted <14 days prior to C1D1.
  * Platelets ≥50,000/ uL. Platelet transfusions are not permitted <14 days prior to C1D1.
  * Hemoglobin ≥ 7 g/dL. RBC transfusions are not permitted <14 days prior to C1D1.
  * Total bilirubin ≤ 1.5 X ULN, or ≤3 x ULN with documented liver metastases and/or Gilbert's Disease
  * AST(SGOT)/ALT(SGPT) ≤2.5 × institutional upper limit of normal, or ≤5 X ULN with documented liver metastases
  * Creatinine clearance ≥ 30 ml/min using Cockcroft/Gault formula
* Able to adhere to the study visit schedule and other protocol requirements.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Prior treatment with CD19 targeted therapy.
* Participants who are receiving any other investigational agents.
* Clinically significant third space fluid accumulation (i.e., ascites requiring drainage or pleural effusion that is either requiring drainage or associated with shortness of breath) unless proven by cytology to be malignant due to WM.
* Pregnant or breastfeeding.
* Participants with known CNS lymphoma.
* Participants with known history of Human Immunodeficiency Virus (HIV), chronic hepatitis B virus (HBV) or hepatitis C (HCV) requiring active treatment. Note: Participants with serologic evidence of prior vaccination to HBV (i.e., HBs Ag-, and anti-HBs+ and anti-HBC-) and positive anti-HBc from IVIG may participate.
* Significant cardiovascular disease defined as:

  * Unstable angina within the past 6 months, or
  * History of myocardial infarction within the past 6 months
  * Any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification, or
  * Uncontrolled or symptomatic arrhythmias
* Participants with a history of Stevens-Johnson syndrome (SJS) or Toxic Epidermal Necrolysis (TEN)
* Concurrent systemic immunosuppressant therapy.
* Vaccinated with live, attenuated vaccines within 4 weeks of first dose of study drug.
* Recent infection requiring systemic treatment that was completed ≤ 14 days before the first dose of the study drug.
* Major surgery within 4 weeks of first dose of study drug.
* Participants with ongoing alcohol or drug abuse.
* History of a non-lymphoma malignancy, except adequately treated local basal cell or squamous cell carcinoma of the skin, cervical carcinoma in situ, superficial bladder cancer, localized prostate cancer, other adequately treated stage 1 or 2 cancer currently in complete remission, or any other cancer that is in a complete remission.
* Prior or ongoing clinically significant illness, medical condition, surgical history, physical finding, EKG finding, or laboratory abnormality that, in the investigator's opinion, could affect the safety of the patient; alter the absorption, distribution, metabolism or excretion of the study drug; or impair the assessment of study results.
* Participants with ongoing >grade 1 toxicities from prior therapy (alopecia any grade and/or grade 2 neuropathy are permitted).
* Participants with clinically significant history of liver disease, including cirrhosis or hepatitis (viral, autoimmune, etc).
* Participants who are unwilling or unable to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-02-17 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | 4 weeks up to 6 months
  Overall Response Rate= Minor response (>25%-50% reduction in serum IgM from baseline) + Partial Response (>50-90% reduction in serum IgM from baseline) + Very Good Partial Response (>90% reduction in serum IgM from baseline) + Complete Response (resolution of all symptoms, normalization of serum IgM with disappearance of IgM paraprotein, resolution of any adenopathy or splenomegaly).

SECONDARY OUTCOMES:
Number of Participants With Complete Response | 6 months
  A complete response is defined as having resolution of WM related symptoms, normalization of serum IgM levels with complete disappearance of IgM paraprotein by immunofixation, and resolution of any adenopathy or splenomegaly.
Number of Participants With Very Good Partial Response | 6 months
  Very Good Partial Response (VGPR): is defined as ≥90% reduction in serum IgM levels, or normalization of serum IgM levels.
Number of Participants With Partial Response | 6 months
  Partial response (PR) is defined as achieving a ≥50% reduction in serum IgM levels.
Number of Participants With Minor Response | 6 months
  Minor Response (MR): A minor response (MR) is defined 25-49% reduction in serum IgM levels.
Number of Participants With Stable Disease | 6 months
  Stable disease is defined as having <25% increase in serum IgM levels and <25% reduction in serum IgM levels
Progression Free Survival | 3 years
  Amount of time following loncastuximab administration until >25% increase in serum IgM
Bone marrow response | 6 months
  Absolute change in bone marrow burden of disease from baseline
Overall Response Rate Among Participants Without MYD88 Mutations | 6 months
  Overall Response Rate in participants who tested negative for a MYD88 mutation= Minor response (>25%-50% reduction in serum IgM from baseline) + Partial Response (>50-90% reduction in serum IgM from baseline) + Very Good Partial Response (>90% reduction in serum IgM from baseline) + Complete Response (resolution of all symptoms, normalization of serum IgM with disappearance of IgM paraprotein, resolution of any adenopathy or splenomegaly).
Overall Response Rate Among Participants Without CXCR4 Mutations | 6 months
  Overall Response Rate in participants who tested negative for a CXCR4 mutation= Minor response (>25%-50% reduction in serum IgM from baseline) + Partial Response (>50-90% reduction in serum IgM from baseline) + Very Good Partial Response (>90% reduction in serum IgM from baseline) + Complete Response (resolution of all symptoms, normalization of serum IgM with disappearance of IgM paraprotein, resolution of any adenopathy or splenomegaly).
Number of Participants With Treatment-related Adverse Events | 6 months
  Number of participants who experienced an adverse event while on loncastuximab tesirine
Number of Participants With IgM Flare | 6 months
  Number of participants who experienced an IgM Flare while on loncastuximab tesirine
Number of Participants With Tumor Lysis Syndrome | 6 months
  Number of participants who experienced Tumor Lysis Syndrome while on loncastuximab tesirine
Impact of loncastuximab tesirine in the participants' quality of life | 6 months
  Quality of life questionnaire European Organisation for Research and Treatment of Cancer. Scores range from 0-100 with high scores indicating a better outcome.
Overall Response Rate Among CXCR4 Mutated Participants | 6 months
  Overall Response Rate for participants who tested positive for a CXCR4 mutation= Minor response (>25%-50% reduction in serum IgM from baseline) + Partial Response (>50-90% reduction in serum IgM from baseline) + Very Good Partial Response (>90% reduction in serum IgM from baseline) + Complete Response (resolution of all symptoms, normalization of serum IgM with disappearance of IgM paraprotein, resolution of any adenopathy or splenomegaly).
Overall Response Rate Among Participants With MYD88 Mutations | 6 months
  Overall Response Rate in participants who tested positive for a MYD88 mutation= Minor response (>25%-50% reduction in serum IgM from baseline) + Partial Response (>50-90% reduction in serum IgM from baseline) + Very Good Partial Response (>90% reduction in serum IgM from baseline) + Complete Response (resolution of all symptoms, normalization of serum IgM with disappearance of IgM paraprotein, resolution of any adenopathy or splenomegaly).

CONTACTS AND LOCATIONS:
Overall Officials: Shayna Sarosiek, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Fred Hutch, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu